CLINICAL TRIAL: NCT01786577
Title: Neuroimaging Biomarkers for Post-Operative Cognitive Decline in Older Adults
Brief Title: Study To Analyze Memory/Thinking Problems In Older Adults After Surgery
Acronym: POCD
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201601040-N; R01NR014181-01 (NIH); 487-2012 (Other: UF legacy)
Record Dates: First submitted 2013-01-30; First posted 2013-02-08 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Post-Operative Cognitive Decline in Older Adults
Keywords: Neuroimaging Biomarkers; Cognitive Decline in Elderly; Memory, Thinking problems for Older Adults; Executive Decline; Post-operative cognitive change
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgery: 80 patients will undergo total knee replacement surgery; two Magnetic Resonance Imaging scans; cognitive assessment testing.
  Interventions: Other: Magnetic Resonance Imaging; Behavioral: Cognitive assessment testing
- Non-Surgery: 80 non-surgery participants will be included as part of the control group; two Magnetic Resonance Imaging scans; cognitive assessment testing.
  Interventions: Other: Magnetic Resonance Imaging; Behavioral: Cognitive assessment testing

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Both groups will undergo two MRIs at baseline and within 48 hours after surgery/non-surgery.
  Other Names: MRI
Behavioral: Cognitive assessment testing — Both groups will undergo in-person baseline assessment of cognitive functioning as well as assessments at three weeks, three months and one year.
  Other Names: Cognitive assessement tests

SUMMARY:
The purpose of the study is to examine specific neuroimaging predictors of memory and executive decline in older adults at various stages after total knee replacement surgery.

DETAILED DESCRIPTION:
Cognitive impairment after major cardiac or non-cardiac surgery occurs in a high rate for older adults. The results of previous studies indicate that certain neuro-imaging markers can determine which individuals pose a greater risk for memory and thinking changes after surgery. Based on a pilot study, there is evidence that pre-surgical neuroimaging biomarkers associate with memory and executive decline after a well controlled surgical procedure (total knee antroplasty). In this study, researchers will use brain imaging studies to determine which patients are most likely to be affected by cognitive changes after this type of surgery. The use of Magnetic Resonance Imaging (MRI) will help investigators identify brain biomarkers that are associated with cognitive problems, such as white matter abnormalities and changes to small blood vessels. Patients undergoing total knee replacement surgery, as well as a group of non-surgery participants of similar age, education and health status,will receive cognitive testing and MRI brain scans before and after surgery/non-surgery. Researchers will compare and monitor both groups up to one year after surgery/non-surgery.

Prior to enrollment, participants will be asked to review the informed consent and provide written consent to participate in the study. The enrollment phase will involve in-person baseline assessment of cognitive functioning within two weeks of the scheduled surgery/non-surgery in order to rule out exclusion criteria. Testing will be in cooperation with the University of Florida General Clinical Research Center. Post-baseline MRI will be conducted on all participants (surgery/control) within 48 hours of the surgery/pseudo-surgery date to identify acute stroke differences from baseline. Cognitive assessments will be conducted for each participant at three-weeks, three-months, and one-year after surgery.

The research is highly significant because it will be the first study to use in-vivo diffusion imaging methods to examine the contribution of specific presurgical neuroanatomical vulnerabilities on executive and memory cognitive decline after one of the most common orthopedic surgeries sought by older adults. Additionally, it will be the first study to examine how specific neuroimaging biomarkers interact negatively with specific peri-operative variables including emboli number during surgery, embolic changes to the brain, anesthesia depth, and cerebral oxygenation.

The findings of the study will improve pre-surgery screening procedures for older adults and assist with the development of peri-operative interventions that will prevent neurodegenerative disease acceleration.

ELIGIBILITY:
Inclusion Criteria:

* Planned total unilateral knee antroplasty or non-surgical knee osteoarthritis
* Age 60 years or older at the time of baseline assessment
* Telephone screening and in-person baseline cognitive testing not supportive of dementia
* Handedness: Right handed; restriction to left-right hemisphere laterality and white matter pathways
* Participant and family deny presence of difficulties with Instrumental Activities of Daily Living (IADL)
* All ethnic and racial groups will be recruited

Exclusion Criteria:

* Underlying medical diseases likely to limit lifespan or confound outcome analyses:

  1. cancer requiring treatment in past five years
  2. serious infectious diseases
  3. congestive heart failure
  4. chronic hepatitis
  5. history of organ transplantation
  6. seizure disorders
  7. history of head trauma resulting in intensive care
  8. current diagnosis of alcoholism, drug dependence, history of major tranquilizer use
* Neurodegenerative Exclusions:

  1. history of major stroke
  2. exposure to toxins or neuroleptics
  3. history of encephalitis
  4. neurological signs of upper motor neuron disease, cerebellar involvement, supranuclear palsy, or significant orthostatic hypertension
  5. signs of dementia.
* Psychiatric Exclusions:

  1. major psychiatric disorder
  2. major depression
* Conditions or behaviors likely to affect imaging or cognitive testing:

  1. claustrophobia
  2. non-medical bodily metal, pace-maker device
  3. less than five years of formal education
  4. inability to read or write
  5. self-reported hearing difficulty that interferes with standardized test administration

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two age-matched participant groups will be recruited. Healthy non-demented age matched patients undergoing elective total knee arthoplasty, and age, education, and diseased matched (osteoarthritis knee pain;) non-surgery peers.
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2013-03-19 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
Predicting Executive Decline | baseline, 3 weeks, 3 months, 1 year
  Severity of pre-surgical/baseline neuroimaging markers of cerebrovascular disease will predict post-operative executive decline at 3 weeks, 3 months and 1 year.
Predicting Memory Decline | baseline, 3 weeks, 3 months, 1 year
  Pre-surgical/baseline neuroimaging markers of entorhinal-hippocampal white matter connectivity will predict post-operative memory decline at 3 weeks, 3 months and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Price, Ph.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Hizel LP, Warner ED, Wiggins ME, Tanner JJ, Parvataneni H, Davis R, Penney DL, Libon DJ, Tighe P, Garvan CW, Price CC. Clock Drawing Performance Slows for Older Adults After Total Knee Replacement Surgery. Anesth Analg. 2019 Jul;129(1):212-219. doi: 10.1213/ANE.0000000000003735. PMID 30273231